CLINICAL TRIAL: NCT02871674
Title: Good Night Project: Behavioural Sleep Interventions for Children With ADHD: A Randomised Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Leeds (Other)
Collaborators: Shaqra University (Other)
Responsible Party: Principal Investigator, Hetaf Alammar, PhD student, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000
Record Dates: First submitted 2016-08-09; First posted 2016-08-18 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Attention Deficit Hyperactivity Disorders; Neurodevelopmental Disorders; Attention Deficit Disorder With Hyperactivity
Keywords: Behavioural interventions; Sleep difficulties; Children; Attention Deficit Hyperactivity Disorder; Randomised controlled trial; Saudi Arabia; Behavioural Insomnia
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will receive behavioural training by psychologists in three sessions over three weeks
  Interventions: Behavioral: Good Night Project
- Control group - usual care (No Intervention): Participants in the control group will receive usual care. They will also attend their usual appointments with the psychiatrists. They will not receive any intervention.

INTERVENTIONS:
Behavioral: Good Night Project — The behavioural interventions have been designed on the basis of three sources. Firstly, a systematic review conducted by the research team that examined the best evidence in the field in different countries. Secondly, a Delphi study, which aimed to identify behavioural interventions that can be used to manage sleep difficulties in Saudi Arabia in accordance with professionals' views and primary caregivers' needs, and which was also conducted by the research team. Thirdly, evidence-based practice resources that help in understanding and managing sleep difficulties will be translated into Arabic.
  Arms: Intervention group

SUMMARY:
The study aims to implement and evaluate an RCT of behavioural sleep interventions for children aged 5-12 years with ADHD, and their primary caregivers, (women) in Saudi Arabia to address the following questions:

1. To what extent can a behavioural intervention improve sleep difficulties and increase sleep duration in children with ADHD?
2. To what extent do intervention-induced changes in sleep for children or primary caregivers (women) account for any changes in ADHD symptoms?

ELIGIBILITY:
Inclusion Criteria:

* The participants will be primary caregivers (women) of children aged 5-12 years who have been diagnosed with ADHD by a psychiatrist, using the criteria taken from Diagnostic and Statistical Manual of Mental Disorders-5 in Saudi Arabia.
* Children with comorbidities will be also included.
* Sleep difficulties are defined as a total score of over 41 in the Children's Sleep Habits Questionnaire (CSHQ).

Exclusion Criteria:

Children will be excluded from the study if they meet any of the following criteria:

* They receive non-pharmacological interventions for their sleep difficulties.
* They have been previously diagnosed as having an intellectual disability (IQ < 70).
* They have obstructive sleep apnoea, according to the three items in the CSHQ.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
The Children's Sleep Habits Questionnaire CSHQ | 2 months
  This is used widely to assess sleep, pre and post intervention, and focuses on measurement of the following subscales: Bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night waking, parasomnias, sleep-disordered breathing and daytime sleepiness. Higher scores indicate significant sleep difficulties.
Conners' Parent Rating Scale-48 (CPRS-48) | 2 months
  This scale consists of 48 items that focus on five subscales: conduct problems, learning disabilities, psychosomatic disorders, impulsivity and hyperactivity and anxiety. It focuses on children aged 3-17 years.

SECONDARY OUTCOMES:
The Sleep Disorders Scale for primary caregivers | 2 months
  This scale consists of 36 items that focus on sleep difficulties in adults, and is divided according to the following subscales: insomnia, hypersomnia, circadian rhythm sleep disorders, sleep terrors and sleepwalking.
The Depression Anxiety Stress Scales DASS | 2 months
  This is designed to measure negative emotions in adults, according to three subscales: depression, anxiety and stress.
Conners' Teachers Rating Scale-28 (CTRS-28) | 1 month
  This scale consists of 28 items that focus on three subscales: Conduct problems, Hyperactivity, Inattentive and Passive. It focuses on children aged 3-17 years.

OTHER OUTCOMES:
Activity monitor (ActiGraph) | 1 month
  This outcome records the physical activity in order to provide sleep duration in seven days at baseline and seven days after a month of randomization to measure change. It will be used as an objective measure with some participants.
Activity monitor diary | 1 month
  This outcome records sleep/wake time and related information in seven days at baseline and seven days after a month of randomization to measure change. It will be used with some participants to support Activity monitor (ActiGraph) measure.
Demographic form | Baseline
  The form will be used to collect demographic information for both primary caregivers and their children

CONTACTS AND LOCATIONS:
Overall Officials: Hetaf A Alammar, PhD student, Principal Investigator — University of Leeds